CLINICAL TRIAL: NCT02337192
Title: Oral Decontamination Using Antimicrobial Photodynamic Therapy Applied in Orthodontic Patients.
Brief Title: Antimicrobial Photodynamic Therapy Applied in Orthodontic. Orthodontic Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fernanda Rossi Paolillo, Vitor Hugo Panhóca, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: orto14
Record Dates: First submitted 2014-12-04; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Dentist-Patient Relations
Keywords: Orthodontic, Photochemoterapy
MeSH Terms: interventions — Curcumin; TBP1901; Surface-Active Agents; Dimethyl Sulfoxide; Water; chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group 1 (Experimental): Negative control - Moutwash with 1,5mL of dimethyl sulfoxide at 5% (DMSO) in water solution - During 2 minutes.
  Interventions: Drug: DMSO + water
- Group 2 (Experimental): Mouthwash with Swish with Curcumin
  Interventions: Drug: Curcumin
- Group 3 (Experimental): Moutwash with Swish with Curcumin + SDS
  Interventions: Drug: Curcumin; Drug: Surfactant
- Group 4 (Experimental): Experiment use dental irradiation with blue light (LED) only.
  Interventions: Device: LED
- Group 5 (Experimental): Antimicrobial Photodynamic Therapy (APDT) with blue light and Curcumin salt.
  Interventions: Drug: Curcumin; Device: LED
- Group 6 (Experimental): Antimicrobial Photodynamic Therapy (APDT) with blue light, Curcumin salt and surfactant.
  Interventions: Drug: Curcumin; Device: LED; Drug: Surfactant
- Group 7 (Experimental): Positive control - Use of mouthwash with Chlorhexidine only
  Interventions: Drug: Chlorhexidine gluconate

INTERVENTIONS:
Drug: Curcumin
  Other Names: Curcumin salt
  Arms: Group 2; Group 3; Group 5; Group 6
Device: LED
  Arms: Group 4; Group 5; Group 6
Drug: Surfactant
  Arms: Group 3; Group 6
Drug: DMSO + water
  Arms: Group 1
Drug: Chlorhexidine gluconate
  Arms: Group 7

SUMMARY:
We demonstrated the use of the Antimicrobial Photodynamic Therapy as a coadjutant oral decontamination agent. It was also shown that SDS surfactant improves the antibacterial action of APDT when using Curcumin as the photosensitizer. The decontamination levels obtained with APDT are comparable with the levels observed with the use of Chlorhexidine. The clinical relevancy is the control of oral microbial load which will improve the patients' quality of life and will decrease the possibility of cross contamination in the dental office.

DETAILED DESCRIPTION:
The installation of the orthodontic appliances promotes an increase in the retentive area available for microbial aggregation, difficult the oral health promotion and, in addition, promotes the artificial selection of biofilms containing a higher load of pathogenic microorganisms. In this way, it becomes of critical importance, the development of techniques that might aid in the reduction of the oral microbial load. One possible approach is the use of the Antimicrobial Photodynamic Therapy (APDT). In this direction, the objective of this study was to assess the clinical utility of the APDT and the association of the APDT with the SDS surfactant as oral decontamination agents in orthodontic patients. The selected patients (n=24) were randomly distributed within seven experimental groups: G1 - Negative control, G2 - Curcumin mouthwash, G3 - Curcumin mouthwash+SDS, G4 - light irradiation, G5 - APDT, G6 - APDT+SDS and G7 - Positive Control (Chlorhexidine mouthwash). Nonstimulated saliva samples were collected from each one of the patients in three steps (S), as follows: S1- Initial condition, S2 - Treatment with mouthwashes (water, Chlorhexidine or Curcumin) and S3 - After APDT treatment. The efficacy of the proposed treatment protocols was assessed in function of the survival fraction observed in each group. The obtained results were statistically analyzed using variance analysis (ANOVA) and the Kruskal-Wallis test.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were: being under fixed orthodontic treatment, absence of clinical signs of periodontal disease, not used antibiotics 90 days prior to the participation on this study and not use fluoride mouthwashes.

Exclusion Criteria:

* Exclusion criteria were: signs of uncontrolled systemic diseases (diabetes, high blood pressure and heart conditions), breast feeding or pregnant women, patients with oral tumors and patients with history of allergy to any of the materials used, such as Curcumin and Chlorhexidine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Microbiological analysis by the total number of colony-forming units (CFU) | one section ( one hour)

CONTACTS AND LOCATIONS:
Overall Officials: Vitor H Panhóca, Ms, Principal Investigator — University of Sao Paulo
Locations (1):
- Vitor Hugo Panhóca, São Carlos, São Paulo, Brazil

REFERENCES:
- [Result] Iliadi A, Baumgartner S, Athanasiou AE, Eliades T, Eliades G. Effect of intraoral aging on the setting status of resin composite and glass ionomer orthodontic adhesives. Am J Orthod Dentofacial Orthop. 2014 Apr;145(4):425-33. doi: 10.1016/j.ajodo.2013.11.020. PMID 24703280